CLINICAL TRIAL: NCT00006176
Title: Clinical, Molecular and Biochemical Characterization of Familial Encephalopathy With Neuroserpin Inclusion Bodies
Brief Title: Clinical and Genetic Studies of Familial Presenile Dementia With Neuronal Inclusion Bodies
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000191; 00-HG-0191
Record Dates: First submitted 2000-08-12; First posted 2000-08-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-04

CONDITIONS: Familial Dementia With Neuroserpin Inclusion Bodies; Nervous System Heredodegenerative Disorder
Keywords: FENIB; Presenile Dementia; Progressive Myoclonic Epilepsy; Dementia; Early Onset Progressive Dementia; Familial Presenile Dementia; FDNIB; familial encephalopathy with neuroserpin inclusion bodies; Heredodegenerative Disorders, Nervous System
MeSH Terms: conditions — Familial encephalopathy with neuroserpin inclusion bodies; Heredodegenerative Disorders, Nervous System; Alzheimer Disease; Myoclonic Epilepsies, Progressive; Dementia

SUMMARY:
The purpose of this study is to learn more about the medical problems and the genetic factors involved in a recently defined form of inherited dementia called "familial dementia with neuroserpin inclusion bodies (FDNIB)." Abnormal substances in nerve cells of patients with this disease affect brain and nervous system function, causing confusion, memory decline and impaired cognition (thinking ability). Patients also develop movement disorders and, possibly, seizures. Symptoms begin in midlife, between 45 and 55 years of age.

Patients with FDNIB and family members 18 years of age or older at risk for the disease may be eligible for this 3-year study.

Participants will have a medical and family history and review of medical records; interview with a medical geneticist (specialist in genetics); physical, neurological and psychiatric examinations; and the following tests and procedures:

1. Blood tests to assess general health
2. Chest and skull X-rays
3. Electrocardiogram (EKG)-record of the electrical activity of the heart using electrodes placed on the chest
4. Electroencephalogram (EEG)-record of the electrical activity of the brain using electrodes placed on the head
5. Ultrasound of the abdomen-imaging of abdominal organs using sound waves
6. Brain magnetic resonance imaging (MRI)-imaging of the brain using a strong magnetic field and radio waves
7. Hearing evaluation
8. Assessment of performance of daily living activities
9. Single photon emission computed tomography (SPECT)-imaging of brain metabolism and blood flow using a radioactive substance injected into a vein

The evaluation will be done over a 3- to 4-day period. At their completion, participants will meet with a physician and a genetics counselor to discuss the clinically significant findings. Participants may be asked to return for follow-up evaluations every 6 months to a year (depending on the individual's condition) for 3 years.

DETAILED DESCRIPTION:
This project involves the study of a novel familial neurodegenerative disorder, familial encephalopathy with neuroserpin inclusion bodies (FENIB). This disorder, which has a characteristic clinical course of progressive dementia and neurologic involvement, was initially defined in one extended family. Neuroserpin is the gene for this disorder and a mutation is present in this large kindred and four additional families/cases. This protocol will characterize the clinical phenotype, delineate the natural history of the disorder and explore genotype/phenotype correlations in the index family and possibly in other reported cases. Families with immunohistopathologically-neuroserpin positive neuronal inclusions on autopsy/biopsy in an affected member(s), neuroserpin mutation-positive proband, or with familial presenile dementia with neurologic features consistent with the original FENIB family will be enrolled.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with a family history of early-onset progressive dementia or decline in cognition and neuronal inclusion bodies which are immunohistopathologically consistent with neuroserpin inclusion bodies.

Children with progressive dementia and myoclonic epilepsy which is consistent with the reported clinical course in pediatric patients or children with the clinical phenotype who on autopsy demonstrate neuronal inclusion boidies which are immunohistopathologically consistent with neuroserpin inclusion bodies.

Family members at risk, of at least 18 years of age, including first degree relatives of affected patients and the adult offspring of these first degree relatives.

In rare instances probands and their at risk family members with known presenile dementia and a neurologic course typical of that seen in FENIB will be enrolled.

We may also enroll offsite individuals who have any of the above findings, but are too medically fragile to travel to the Clinical Center and for whom a durable power of attorney (DPA) is available. The physical examination and laboratory research studies will be performed by the Investigator(s) and all clinical studies will be done in a local accredited hospital.

Family members either not at risk and unaffected spouses may enroll primarily for genetic linkage information. These individuals will contribute a blood sample for molecular analysis only. Those unwilling to travel may also provide a blood sample only. No clinical studies will be performed on individuals from this category.

EXCLUSION CRITERIA:

Another diagnosis of presenile demential is made by a physician including but not limited to: 1) Huntington Disease, 2) Parkinson Disease/Diffuse Lewy Body Disease, 3) Familial Alzheimer Disease with known mutations in presenilin 1, presenilin 2 or beta-amyloid precursor protein, 4) Lafora Body Disease, 5) Pick's Disease, and 6) fronto-temporal dementia.

A Durable Power of Attorney is not available in a human subject that is not medically competent to give consent.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2000-08-10; Primary Completion 2009-08-04 (Actual); Study Completion 2009-08-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Davis RL, Shrimpton AE, Holohan PD, Bradshaw C, Feiglin D, Collins GH, Sonderegger P, Kinter J, Becker LM, Lacbawan F, Krasnewich D, Muenke M, Lawrence DA, Yerby MS, Shaw CM, Gooptu B, Elliott PR, Finch JT, Carrell RW, Lomas DA. Familial dementia caused by polymerization of mutant neuroserpin. Nature. 1999 Sep 23;401(6751):376-9. doi: 10.1038/43894. PMID 10517635
- [Background] Davis RL, Shrimpton AE, Carrell RW, Lomas DA, Gerhard L, Baumann B, Lawrence DA, Yepes M, Kim TS, Ghetti B, Piccardo P, Takao M, Lacbawan F, Muenke M, Sifers RN, Bradshaw CB, Kent PF, Collins GH, Larocca D, Holohan PD. Association between conformational mutations in neuroserpin and onset and severity of dementia. Lancet. 2002 Jun 29;359(9325):2242-7. doi: 10.1016/S0140-6736(02)09293-0. PMID 12103288
- [Background] Davis RL, Holohan PD, Shrimpton AE, Tatum AH, Daucher J, Collins GH, Todd R, Bradshaw C, Kent P, Feiglin D, Rosenbaum A, Yerby MS, Shaw CM, Lacbawan F, Lawrence DA. Familial encephalopathy with neuroserpin inclusion bodies. Am J Pathol. 1999 Dec;155(6):1901-13. doi: 10.1016/S0002-9440(10)65510-1. PMID 10595921